CLINICAL TRIAL: NCT06041724
Title: Single-arm II Phase Study of Envafolimab Combined With Recombinant Human Endostatin and First-line Chemotherapy
Brief Title: Envafolimab Combined With Recombinant Human Endostatin and First-line Chemotherapy Treat of Advanced Mucosal Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Professor and Chief Surgeon, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan-MM003
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Advanced Mucosal Melanoma
MeSH Terms: interventions — Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab combined with recombinant human endostatin and first-line chemotherapy (Experimental)
  Interventions: Drug: Envafolimab combined with recombinant human endostatin and first-line chemotherapy

INTERVENTIONS:
Drug: Envafolimab combined with recombinant human endostatin and first-line chemotherapy — Envafolimab: 300mg day1, s.c. Q3W; Recombinant human endostatin: 210mg day1, Intravenous pump for 72 hours, Q3W; Temozolomide: 150 mg/m2 d1-5, i.v. Q3W; Cisplatin: 25 mg/m2 d1-3, i.v. Q3W.
  All of the above drugs were used for 6 cycles, and then Envafolimab and recombinant human endostatin continued only in patients with no progression in the first stage until disease progression as defined by RECIST1.1, unacceptable toxicity, withdrawal from the study or death, or no more than 2 years.

SUMMARY:
This is a phase II, open, single-center study to explore the efficacy and safety of Envafolimab combined with recombinant human endostatin, temozolomide and cisplatin in the treatment of mucosal melanin. At the same time, the tissue and peripheral blood samples of the patients were taken for the determination of PD-L1 expression, ctDNA and other biomarkers and the results were analyzed to find the predictive factors of prognosis or curative effect. Patients with advanced mucosal melanoma who met the inclusion criteria but did not meet the exclusion criteria were enrolled in this study and received 6 cycles of Envafolimab combined with recombinant human endostatin, temozolomide and cisplatin. Patients without progression were then maintained with Envafolimab combined with recombinant human endostatin until disease progression, intolerable adverse reactions, patient death or withdrawal of informed consent. The longest administration time of recombinant human endostatin was no more than 1 year, and that of Envafolimab was not more than 2 years. The efficacy was evaluated for the first time at 6 weeks, every 6 weeks for the following year, and then every 12 weeks until the end of progress or treatment. The examination method was consistent with the baseline; it was expected to be included in the group for 18 months, and clinical observation until disease progression and patient death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender.
* Histology and pathology confirmed advanced mucosal melanoma.
* Gene mutation state is not limited, except BRAFV600 mutation.
* Has not received first-line treatment for advanced melanoma, and temozolomide and cisplatin have been used in the adjuvant therapy phase, except that the adjuvant therapy phase has been over 6 months or more.
* Eastern Cancer Cooperation Group (ECOG) physical condition score (PS) 0-1.
* The estimated survival time is more than 3 months.
* Within 7 days before screening (including 7 days), the laboratory data were required as follows: neutrophil count ≥ 1.5 × 109 shock L, platelet count ≥ 90 × 109 shock L, hemoglobin ≥ 90g/L (no blood transfusion within 14 days), serum total bilirubin ≤ 1.25x normal upper limit (ULN), ALT and AST ≤ 2.5xULN (patients with liver metastasis ≤ 5xULN); serum creatinine ≤ 1.25xULN.
* Have at least one measurable focus (RECIST1.1 standard).
* Subjects (or their legal representatives / guardians) must sign an informed consent form indicating that they understand the purpose of the study, understand the necessary procedures for the study, and are willing to participate in the study.

Exclusion Criteria:

* Patients who have previously used PD-L1 inhibitors, except those who progressed 1 year after the end of adjuvant therapy of PD-L1 monoclonal antibody;
* Allergic to Envafolimab or recombinant human endostatin and experimental chemotherapeutic drugs;
* Received any experimental drugs or antineoplastic drugs within 4 weeks before entering the group;
* There is a risk of bleeding, bleeding events of clinical significance or other taboos in the use of antivascular drugs;
* There is a history of other tumors in the past five years, except for cured cervical cancer or skin basal cell carcinoma;
* There are tumor emergencies that require immediate radiotherapy, such as symptomatic brain or meningeal metastasis, bone-related events, etc;
* Pregnant or lactating women; Fertile women who do not use adequate contraception;
* Alcohol or drug addiction;
* Patients with active, or history of autoimmune diseases that may recur (e.g. systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or patients at high risk (such as immunosuppressive therapy required for organ transplants). Except for autoimmune hypothyroidism that requires only hormone replacement therapy or skin diseases that do not require systemic treatment;
* Patients who need to receive systemic corticosteroids (dose equivalent to > 10mg prednisone / day) or other immunosuppressive drugs within 14 days before enrollment or during the study. The use of topical or inhaled corticosteroids, or short-term (≤ 7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune and infrequent allergic diseases;
* Important organ failure or other serious diseases, including interstitial pneumonia, clinically related coronary artery disease, cardiovascular disease or myocardial infarction, congestive heart failure, unstable angina pectoris, symptomatic pericardial effusion or unstable arrhythmia within 6 months before admission;
* A history of human immunodeficiency virus infection, or other acquired, congenital immunodeficiency diseases, or a history of organ transplant or stem cell transplantation;
* Patients with active chronic hepatitis B or active hepatitis C. HBV carriers, stable hepatitis B (DNA titer ≤ 103copies / ml) and cured hepatitis C patients (HCVRNA negative) can be enrolled in the group;
* A history of severe neurological or psychiatric illness; severe infection; active disseminated intravascular coagulation or other concomitant diseases that, in the opinion of the researchers, seriously endanger the safety of patients or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2025-09-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 12 months
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with measurable lesions achieving a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) criteria.
Disease Control Rate (DCR) | 12 months
  The proportion of participants who achieves a best overall response of CR, PR or stable disease(SD).
Duration of Response (DoR) | 12 months
  The time from the date that response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Overall Survival (OS) | 12 months
  OS is defined as the time from enrollment to death from any cause.
PD-L1 expression from the tissue and peripheral blood samples of the patients | baseline (When entering the group)
  The tissue and peripheral blood samples of the patients were taken for the determination of PD-L1 expression, and the results were analyzed to find the predictive factors of prognosis or curative effect.
ctDNA expression from the tissue and peripheral blood samples of the patients | baseline (When entering the group)
  The tissue and peripheral blood samples of the patients were taken for the determination of ctDNA expression, and the results were analyzed to find the predictive factors of prognosis or curative effect.
Adverse Events (AEs) according to CTCAE v5.0. | 12 months
  Adverse Events (AEs) according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Luo, M.D, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No